CLINICAL TRIAL: NCT00551564
Title: A Single-Center, Non-Randomized, Open-Label, Comparative Study to Assess the Utility of Novel Technologies and Biomarkers as Methods for Measuring Human Pharmacodynamic Response to 8 Weeks of Administration of Rosiglitazone Maleate 4mg BID in Healthy Normal or Overweight Controls, Healthy Obese Subjects and Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Study to Determine the Utility of Novel Technologies and Biomarkers to Measure Human Response to Rosiglitazone Maleate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DIX110434
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: total body water; T2DM,; Healthy Obese,; Insulin Resistance,; Rosiglitazone maleate,; Glucose Disposal,; hyperinsulinemic-euglycemic clamp,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects in healthy normal and overweight control arm (Experimental): Subjects in the Healthy Normal or Overweight Control Population will be included in this arm and they will receive Rosiglitazone 4 milligram twice daily.
  Interventions: Drug: rosiglitazone maleate
- Subjects in healthy obese with T2DM arm (Experimental): Subjects who are in the Healthy Obese or T2DM Population will be included in this arm and they will receive Rosiglitazone 4 milligram twice daily.
  Interventions: Drug: rosiglitazone maleate

INTERVENTIONS:
Drug: rosiglitazone maleate — Rosiglitazone tablets 4 mg dose will be administered orally by subjects

SUMMARY:
Insulin resistance (IR) is common in many metabolic disorders and predisposes an individual to Type 2 Diabetes Mellitus (T2DM), the Metabolic Syndrome and coronary atherosclerosis. Non-diabetics with IR are at risk, but can be difficult to diagnose.

A major problem with the use of IR as a predictor or marker of disease is the lack of a simple, robust test that can be used to quantify this parameter in a wide variety of clinical situations. The current 'gold standard' methods for measuring insulin sensitivity, such as the hyperinsulinemic-euglycemic (H-E) clamp, are complex, time consuming and costly. Alternative, simpler methods, such as the Homeostasis Model Assessment (HOMA-IR) score, may be less accurate and are not widely accepted.

DETAILED DESCRIPTION:
A Single-Center, Non-Randomized, Open-Label, Comparative Study to Assess the Utility of Novel Technologies and Biomarkers as Methods for Measuring Human Pharmacodynamic Response to 8 Weeks of Administration of Rosiglitazone Maleate 4mg BID in Healthy Normal or Overweight Controls, Healthy Obese Subjects and Subjects with Type 2 Diabetes Mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Male and/or females aged 18-65 years
* Females must either be of non-childbearing potential or childbearing potential (but not pregnant) and using appropriate methods of contraception.
* Healthy normal or overweight control subjects or healthy obese subjects or subjects with T2DM.

Exclusion Criteria:

* Clinically significant past or current medical conditions
* Clinically significant abnormalities in vital signs or routine laboratory parameters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07-31 (Actual); Primary Completion 2008-09-08 (Actual); Study Completion 2008-09-08 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | baseline and after 8 weeks of Rosiglitazone treatment

SECONDARY OUTCOMES:
Insulin resistance | baseline, after 2 weeks treatment, 2 weeks after discontinuation treatment
hepatic glucose output: baseline, after 8 weeks treatment Insulin secretion from oral glucose tolerance | baseline, after 8 weeks treatment
Body composition | baseline & after 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study DIX110434 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/DIX110434?search=study&search_terms=DIX110434#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: DIX110434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register